CLINICAL TRIAL: NCT02923089
Title: The Love of Lentils (LoL) Study - Phase 2: The Effect of Acute Consumption of Lentil-containing Food Products on Post-prandial Blood Glucose and Insulin in Healthy Adults
Brief Title: Postprandial Blood Glucose and Insulin Levels Following Consumption of Lentil-containing Food Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Principal Investigator, Alison Duncan, Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16AU008
Record Dates: First submitted 2016-09-25; First posted 2016-10-04 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Postprandial Glycemia in Healthy Adults
Keywords: Diabetes; Lentils; Pulses; Postprandial glycemia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Small Green Lentil Muffin (Experimental): Muffin: 25g available carbohydrate from small green lentil
  Interventions: Other: Muffin: 25g available carbohydrate from small green lentil
- Split Red Lentil Muffin (Experimental): Muffin: 25g available carbohydrate from split red lentil
  Interventions: Other: Muffin: 25g available carbohydrate from split red lentil
- Wheat Muffin (Placebo Comparator): Muffin: 25g available carbohydrate from wheat
  Interventions: Other: Wheat muffin
- Small Green Lentil Soup (Experimental): Soup: 25g available carbohydrate from small green lentil
  Interventions: Other: Soup: 25g available carbohydrate from small green lentil
- Split Red Lentil Soup (Experimental): Soup: 25g available carbohydrate from split red lentil
  Interventions: Other: Soup: 25g available carbohydrate from split red lentil
- Potato Soup (Placebo Comparator): Soup: 25g available carbohydrate from potato
  Interventions: Other: Potato soup
- Small Green Lentil Chili (Experimental): Chili: 25g available carbohydrate from small green lentil
  Interventions: Other: Chili: 25g available carbohydrate from small green lentil
- Split Red Lentil Chili (Experimental): Chili: 25g available carbohydrate from split red lentil
  Interventions: Other: Chili: 25g available carbohydrate from split red lentil
- Rice Chili (Placebo Comparator): Chili: 25g available carbohydrate from rice
  Interventions: Other: Rice chili

INTERVENTIONS:
Other: Muffin: 25g available carbohydrate from small green lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Small Green Lentil Muffin
Other: Muffin: 25g available carbohydrate from split red lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Split Red Lentil Muffin
Other: Wheat muffin — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Wheat Muffin
Other: Soup: 25g available carbohydrate from small green lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Small Green Lentil Soup
Other: Soup: 25g available carbohydrate from split red lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Split Red Lentil Soup
Other: Potato soup — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Potato Soup
Other: Chili: 25g available carbohydrate from small green lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Small Green Lentil Chili
Other: Chili: 25g available carbohydrate from split red lentil — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Split Red Lentil Chili
Other: Rice chili — Comparison of postprandial blood glucose and insulin following consumption of food products with and without lentils.
  Arms: Rice Chili

SUMMARY:
This study will recruit 20 healthy adults (male and female) to complete 9 study visits where they will consume different food products (chili, soup and muffin) with or without lentils incorporated into the them. Blood samples will be obtained by finger prick before and for 2 hours after the meal and analyzed for glucose and insulin.

DETAILED DESCRIPTION:
The purpose of the current study is to determine the effects of lentil-containing food products on postprandial blood glucose and insulin levels in healthy premenopausal women and men aged 18-40 years old.This study will use a randomized crossover design. Participants will complete a series of 9 study visits during which participants will consume 9 study treatment meals consisting of muffins, soup and chilli, with and without lentils. Participants will then have their blood sampled for the following 2 hours by finger prick. Participants will remain seated during the test period. All study visits will occur at the Human Nutraceutical Research Unit and be separated by a washout period of 3-7 days. Throughout the study, it will be asked that participants' lifestyle and physical activity remain unchanged. Participants will be instructed to not start any new dietary approaches, and to not start any new natural health products (unless instructed by a physician).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age 18-40 years (aiming for equal distribution among 18-29, 30-40 years of age)
* BMI 20-30 kg/m2

Exclusion Criteria:

* Diabetes (fasting blood glucose ≥7.0 mmol/L and/or 2hr blood glucose >11.1 mmol/L post-75g OGTT) 1
* Impaired Glucose Tolerance (IGT) (Fasting blood glucose 6.1-6.9 mmol/L and/or 2hr blood glucose 7.8-11.0 mmol/L post-75g OGTT) 1
* Blood pressure >140/90 mm Hg
* Any major medical condition including a history of AIDS or hepatitis
* Medical or surgical event requiring hospitalization within 3 months of randomization
* Any medications except a stable dose (3 months) of oral contraceptives, blood pressure or statin medications
* Natural health products (NHPs) used for glycemic control (all other NHPs okay as long as table for 3 months)
* Tobacco use
* Probiotic supplement use
* Dietary fibre supplement use
* Pulse consumption >4 servings per week
* Food allergy or non-food life threatening allergy
* Alcohol consumption >14 drinks/week or >4 drinks/sitting
* Recent or intended significant weight loss or gain (>4 kg in previous 3 months)
* Elite athletes
* Shift workers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | 2 hours postprandial
Postprandial plasma insulin | 2 hours postprandial

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Duncan, PhD, RD, Principal Investigator — University of Guelph
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No